CLINICAL TRIAL: NCT02259387
Title: Adolescents With Migraine: What's Stress Got To Do With It?
Acronym: Adostress
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 13-3128; UL1TR001082 (NIH)
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hair samples for cortisol.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Children with migraines will be placed into this group.
- Controls: Children without migraines or headaches will be placed into this group.

SUMMARY:
The overall objective of this proposal is to better define the relationship between perceived stress, hair cortisol, and migraine in adolescents. This will be done by creating 2 arms of the study: those with migraines (cases) and those without migraines or headaches (controls). Each arm will answer several of the same questionnaires and have hair cortisol samples taken multiple times over the course of 12 weeks.

DETAILED DESCRIPTION:
The overall objective of this proposal is to better define the relationship between perceived stress, hair cortisol, and migraine in adolescents. Although adolescents most frequently report stress as their migraine trigger, stress measurement and treatment are usually beyond the scope of routine clinical care. Hair cortisol levels may identify stressed adolescents who need structured stress management, as well as provide objective evidence for the medical community, migraineurs (i.e. individuals who experience migraines), and their families, who may be reluctant to accept stress as a migraine factor. The rationale for this research is that scientific validation of an association between stress and migraine will inform future prevention studies in the headache field and potentially identify a stress biomarker for migraine.

This prospective study will enroll 67 adolescents (aged 13-17) with migraine and 33 adolescents without migraine for 12 weeks with the following aims:

Aim 1: Measure the relationship between hair cortisol concentration and perceived stress in adolescents with and without migraine.

Hypothesis: The association between hair cortisol and perceived stress (3 month averages) will be a positive in both adolescents with and without migraine.

Aim 2: Measure the relationship between migraine frequency with perceived stress and hair cortisol concentration in adolescents with migraine.

Hypothesis: The association between migraine frequency with (a) perceived stress and (b) hair cortisol will be positive in adolescents with migraines.

ELIGIBILITY:
Inclusion criteria:

For Cases:

* Diagnosis of Migraine as defined by the ICHD-II
* At least 1 migraine per month

For Controls:

* No diagnosis of Migraine as defined by ICHD-II
* No diagnosis of Primary Headache Disorders as defined by ICHD-II

Exclusion Criteria for Migrainers and Non-migrainers:

* A secondary headache disorder as defined by ICHD-II
* A continuous headache (i.e. 24 hours a day every day)
* An underlying neurological condition such as epilepsy, chiari malformation, or neurocutaneous disorder
* A chronic medical illness including those illnesses that require chronic steroid use such as asthma, cancer or rheumatologic disorders
* Subject has bleached hair in past 3 months.
* Pubertal Tanner stage 1 or 2 (Hair cortisol concentration may depend on developmental stage; 59 Tanner staging will be performed by Dr. Kedia).
* Subject is pregnant or has a positive pregnancy test.
* Present psychiatric disease as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM IV) (e.g. psychosis, bipolar disorder, major depression, generalized anxiety disorder), alcohol or drug dependence, or documented developmental delays or impairments (e.g., autism, cerebral palsy, or mental retardation) that, in the opinion of the site investigator, would interfere with adherence to study requirements or safe participation in the trial
* Any and all other diagnoses or conditions which in the opinion of the primary investigator would prevent the patient from being a suitable candidate for the study or interfere with the medical care needs of the study subject.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population to be sampled is adolescents (13-17 years old) with migraines, both male and female. Migraines are common in the pediatric population with a prevalence as high as 10% in children 5-14 years old,1 and 28% in adolescents 15-19 years old (Split W, 1999).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-09-12 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Correlation between hair cortisol and perceived stress | 12 weeks
  Hair cortisol (a biomarker of stress) will be correlated with perceived stress (as measured by participant-answered questionnaires). We expect a positive correlation.
Correlation between headache frequency, perceived stress, and hair cortisol. | 12 weeks
  Hair cortisol (a biomarker of stress) will be correlated with perceived stress (as measured by participant-answered questionnaires) and headache frequency (as measured by a headache diary, which will measure how many days per month a child has headaches). We expect a positive correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Sita Kedia, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Colorado Children's Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Split W, Neuman W. Epidemiology of migraine among students from randomly selected secondary schools in Lodz. Headache. 1999 Jul-Aug;39(7):494-501. doi: 10.1046/j.1526-4610.1999.3907494.x. PMID 11279934